CLINICAL TRIAL: NCT04242641
Title: An Exploratory Study to Determine the Potential Impact of Parental Attendance at WW on Weight and Behavioural Outcomes in Children
Brief Title: An Exploratory Study to Determine the Potential Impact of Parental Attendance at WW on Weight and Behavioural Outcomes in Children: WWChild
Acronym: WWChild
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid pandemic
Sponsor: University of Leeds (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Maria Bryant, Associate Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MREC 19-0.23
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomised on a 1:1 ratio to either the intervention arm (WW programme) or to the control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the which arm the participants have been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW (formally Weight Watchers) (Experimental): The intervention will consist of engaging with the WW programme for 12 weeks, including weekly attendance at a local WW workshop and access to digital tools. Only the parent will take part in the WW intervention. No modifications will be made to the current WW programme to support child weight loss.
  Interventions: Behavioral: WW
- Control (No Intervention): Participants randomised to the control group will receive no intervention during the 3 month period. Following final data collection control participants will receive 3 month complimentary access to WW.

INTERVENTIONS:
Behavioral: WW — WW is a structured lifestyle modification, weight-loss programme involving a programme for healthy eating, physical activity and positive mindset and support via attendance at local WW workshops and digital tools.
  Arms: WW (formally Weight Watchers)

SUMMARY:
The purpose of the WWChild study is to determine the feasibility of assessing the potential impact of parents attendance at WW on their child's weight status and weight related behaviours. The feasibility study will randomly allocate 60 parent participants to either the WW programme (formally Weight Watchers) or to a control arm. Data will be collected from both parent and child at baseline and at three months to explore changes in weight status and weight related behaviours.

DETAILED DESCRIPTION:
Study objectives:

1. To determine if it is possible to recruit parents who have a BMI ≥25 with children whose BMI is over the 85th percentile and assess the recruitment rate.
2. To assess the acceptability and feasibility of collecting height and weight data from both the parent and child during two assessment visits (baseline and follow-up).
3. To explore trends and variance in outcomes between treatment allocation to support the utility of a future definitive trial and to develop a sample size calculation.
4. To assess the acceptability and sensitivity of secondary outcome measures to evaluate the potential impact of parental attendance at WW on weight related behaviours of the family and child (eg. eating habits and physical activity levels).
5. To test the assumptions in the logic model through which parental participation is assumed to impact on child outcomes (Programme Theory).

WWChild is a randomised feasibility study with an embedded process evaluation, aiming to recruit 60 participants. Participants will be recruited through advertising using relevant channels that will target parents of children of primary school age.

All eligible participants will be registered and allocated to either 3 month programme with WW or to a waiting list control arm. Participants initially randomised to the control arm will receive free access to 3 month programme with WW after follow up data has been collected. Children will not attend the WW sessions.

Screening of participants will take place at multiple time-points. The initial screen will be conducted online by people who are interested in the study (self-referred). Those potentially meeting eligibility criteria will be asked to contact researchers at the Clinical Trials Research Unit by telephone or email, who will provide more information about the study and re-assess eligibility. If potentially eligible and interested, they will be invited to a baseline assessment visit, where eligibility will be confirmed, consent will be obtained, participants will be registered and baseline data will be collected. Participants will also be randomised at the end of this visit.

ELIGIBILITY:
Parent Inclusion Criteria:

1. Male or female ages 18-75 years
2. Body Mass Index (BMI) of 25 to 45 (confirmed at baseline by researcher measurement)
3. Self report need to lose weight. Parent/primary care-giver to a child meeting child eligibility criteria
4. Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by physician, with the exception of multivitamins or other vitamin supplement
5. Willing to follow recommendations required by study protocol (2 appointments), including attending programme workshops and using App if assigned to the WW arm
6. Use of a personal smartphone (iOS 9.0 or Android 4.1 or higher with at least 54MB of available storage for Android or 154 MB for iPhone to accommodate the size of the WW app)
7. Residing within 30 miles of a WW workshop
8. Ability to read, write and speak English at an adequate level to receive the intervention

Child Inclusion Criteria

1. Must be at or over the 85th percentile (confirmed at baseline by researcher measurement)
2. Must be aged between 5 and 11 years at baseline
3. Must live with enrolled parent for the majority of the time

Parent Exclusion Criteria:

1. Membership at WW within the past 12 months.
2. Given birth in the past six months, currently pregnant, or planning on becoming pregnant over the next 3 months.
3. Weight loss of ≥ 5 kg in the previous 6 months.
4. History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months.
5. Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
6. Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg (asked as 'high blood pressure in on-line/telephone screen; confirmed at baseline visit)
7. Currently have type 1 or type II diabetes (pre-diabetes acceptable);
8. Currently have chronic/inflammatory gastrointestinal disorder (irritable bowel syndrome acceptable)
9. Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
10. Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qysmia, Contrave, with the exception of those on a stable dose of SSRIs for at least 6 months
11. Ever had surgical procedure for weight loss.
12. Major surgery within the previous 12 months.
13. Presence of implanted cardiac defibrillator or pacemaker.
14. History of cancer within past 5 years or current treatment for cancer (if skin cancer, past 6 months)
15. Currently have a medical diagnosis of Anorexia Nervosa or Bulimia Nervosa
16. Hospitalisation for psychiatric problems during the past 12 months
17. Planning to relocate in the next 12 months
18. Another member (excluding the enrolled child) of the household is participating in this research study

Child Exclusion Criteria

1. Currently enrolled in any weight loss related programmes
2. Diagnosed with Prader- Willi syndrome, Cushing Syndrome, Hypothyroidism or Hashimoto's Disease.
3. Weight loss of ≥ 5% in the previous 6 months.
4. Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
5. Currently have type 1 or type II diabetes (pre-diabetes acceptable);
6. Currently have chronic/inflammatory gastrointestinal disorder (irritable bowel syndrome acceptable)
7. Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
8. Taking any prescription medication with known effects on appetite or weight.
9. Major surgery within the previous 12 months.
10. Presence of implanted cardiac defibrillator or pacemaker.
11. History of cancer within past 5 years or current treatment for cancer
12. Hospitalisation for psychiatric problems during the past 12 months
13. Another child of the household is participating in this research study

    -

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Recruitment to online screener | Baseline
  Number of individuals that self-refer to the WWChild online screener
Number of eligible participant | Baseline
  The number of eligible parent-child dyads that complete both the online and telephone screening process that determines eligibility.
Number of non eligible participant dyads | Baseline
  The number of dyads that complete both the online and telephone screener who are not eligible
Reason for non-eligibility | Baseline
  The number of participants who are ineligible for each reason for not being included in the study
Number of participant dyads invited to baseline appointment | Baseline
  The total number of participant dyads that are invited to attend a baseline appointment following online and telephone eligibility screening
Number of baseline appointments completed | Baseline
  The total number of participant dyads that complete baseline appointments
Number of follow up appointments completed | 3 month follow up
  The total number of participant dyads that complete a 3 month follow up data collection appointment
Number of withdrawals | 3 month follow up
  The total number of withdrawals from the study
Time point of withdrawal | 3 month follow up
  The time point within the study of withdrawals
Reason for withdrawal | 3 month follow up
  The number of participants that withdraw for each reason
Number of parent height and weights collected | 3 month follow up
  The total number of parent participants that have had both their height and weight measured.
Number of child height and weights collected | 3 month follow up
  The total number of child participants that have had both their height and weight collected
Reason for non-completion of data collection protocol | 3 month follow up
  The total number of participant dyads that have not had all data collected according to the protocol for each reason for non completion
Trial acceptability qualitatively assessed through interviews with participants | 3 month follow up
  Qualitative interviews with parents will assess the acceptability of the study.
Compliance with WW intervention | 3 month follow up
  Intervention attendance and usage of the intervention app will be analysed to measure compliance of intervention
Reasons for participation | 3 month follow up
  Qualitative interviews will be used to explore reasons for participation in the study and potential barriers.
Testing of assumptions of parental attendance having potential to impact on child outcomes | 3 month follow up.
  Qualitative interviews will be used to explore assumptions proposed in the logic model that proposes parental attendance at WW has the potential to impact on child outcomes.

OTHER OUTCOMES:
Difference in child BMI (Weight(kg)/ Height(m)²)z score | Baseline and 3 month follow up
  Difference in BMI (Weight(kg)/Height(m)2) z-score change of child from baseline to follow up between groups randomised to receive WW intervention and group randomised to the control group at 3 month post randomisation.
Differences in weight (kg) change of adult | Baseline and 3 month follow up
  Differences in weight (kg) change of adult from baseline to follow up between intervention and control arm at 3 months post randomisation.
Differences in weight (kg) change of child | Baseline and 3 month follow up
  Differences in weight (kg) change of child from baseline to follow up between intervention and control arm at 3 months post randomisation.
Difference in waist circumference (cm) of adult | Baseline and 3 month follow up
  Difference in waist circumference (cm) of adult from baseline to follow up between intervention and control arm at 3 months post randomisation.
Difference in waist circumference (cm) of child | Baseline and 3 month follow up
  Difference in waist circumference (cm) of child from baseline to follow up between intervention and control arm at 3 months post randomisation.
Fitness (sit to stand test) adult | Baseline and follow up
  Difference in fitness measured by the total number of sit to stands completed in one minute from baseline to follow up between intervention and control arm
Fitness (sit to stand test) child | Baseline and follow up
  Difference in fitness measured by the total number of sit to stands completed in one minute from baseline to follow up between intervention and control arm at 3 months post randomisation
Flexibility (sit and reach) adult | Baseline and follow up
  Difference in flexibility measured by the distance reached during the sit and reach test from baseline to follow up between intervention and control arm at 3 month post randomisation
Flexibility (sit and reach) child | Baseline and follow up
  Difference in flexibility measured by the distance reached during the sit and reach test from baseline to follow up between intervention and control arm at 3 month post randomisation
Parenting self-efficacy (via Dumka PSAM). | Baseline and follow up
  Differences in parent self efficacy score based on the Dumka PSAM from baseline to follow up between intervention and control arm
Family eating behaviours (via Golan Family Eating and Activity Habits Questionnaire). | Baseline and 3 month follow up
  Difference in family eating behaviour scores based on the Golan Family Eating and Activity Habits Questionnaire from baseline to follow up between intervention and control arm.
Self-efficacy of diet and exercise behaviours (Sallis 1988) | Baseline and 3 month follow up
  Difference in parent self efficacy of diet and exercise behaviours from baseline to follow up between intervention and control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bryant, PhD, Principal Investigator — Clinical Trials Research Unit, University of Leeds
Locations (1):
- Clinical Trials Research Unit, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No